CLINICAL TRIAL: NCT04227470
Title: Safety, Tolerability, Pharmacodynamics and Efficacy of HBM9161 Weekly Subcutaneous Administration in Patients With Neuromyelitis Optica Spectrum Disorders (NMOSD) in China
Brief Title: A Study of HBM9161 in NMOSD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 9161.2
Record Dates: First submitted 2019-11-21; First posted 2020-01-13 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: NMO Spectrum Disorder
Keywords: NMOSD
MeSH Terms: conditions — Neuromyelitis Optica | interventions — HBM9161

STUDY DESIGN:
Intervention Model Description: Dose exploration study. Two dose groups (340 mg and 680 mg) were planned, 6 subjects at most for 340 mg group and 6 to 12 subjects for 680mg group. Each subject will only participate in one dose group. Escalation to the next dose level decided by PIs and sponsor after evaluating safety data and PD data for lower dose group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: HBM9161, 340mg (Experimental): HBM 9161 injection, 340mg, weekly administered by subcutaneous for a period of 4 weeks.
  Interventions: Drug: HBM9161 Injection
- Experimental: HBM9161, 680mg (Experimental): HBM 9161 injection, 680mg, weekly administered by subcutaneous for a period of 4 weeks.
  Interventions: Drug: HBM9161 Injection

INTERVENTIONS:
Drug: HBM9161 Injection — Subcutaneous injection; Weekly administered for a period of 4 weeks. All subjects are treated with the testing drug, add on intravenous methylprednisolone (ivMP) with gradually reduce the dose then to oral prednisone. After the administration of the testing drug, if the subject's symptoms get worsen, a rescue therapy need to be adopted as based on Investigator's judgement, the testing drug injection should be discontinued.

SUMMARY:
Primary Objectives:To investigate the safety and tolerability of HBM 9161 in patients with attack of NMOSD in China

DETAILED DESCRIPTION:
This is an open-label, dose exploration study.The investigational drug is HBM9161 injection, and the indication is NMOSD.

HBM9161(HL161BKN) is a human monoclonal antibody. HBM9161 targets the neonatal Fc receptor (FcRn) . By blocking the FcRn IgG-Fc binding site and accelerating the degradation of IgG, it can significantly reduce the total IgG level in blood (including pathological IgG).The serum aquaporin 4 antibody (AQP4-IgG) associated with NMOSD is a pathological IgG, so the combination of standard of care which is intravenous methylprednisolone (ivMP) with HBM9161 is expected to rapidly reduce AQP4-IgG levels.

Two dose groups (340 mg and 680 mg) were planned, and each dose group plans to enroll approximately 6 subjects. All subjects are weekly administered the HBM9161 by subcutaneous injection for a period of 4 weeks, together with standard of care which is of intravenous methylprednisolone (ivMP) by subcutaneous for a period of 4 weeks. The study will investigate the safety, and tolerability, pharmacodynamics and efficacy of HBM 9161 in patients with attack of NMOSD in China.

ELIGIBILITY:
Inclusion Criteria:

1. In visit 1, Male or female aged ≥ 18 years.
2. Patient with NMOSD as defined by 2015 NMOSD diagnostic criteria by IPND (International Panel for NMO Diagnosis).
3. Core clinical manifestations characterized by new acute optic neuritis and/or transverse myelitis. A clinical event is defined as an episode of inflammation in the spinal cord and/or optic nerve leading to neurologic deficits which can be identified by physical examination and not attributable to another disease process.
4. The EDSS score should be ≥ 2.5 and ≤7.5 at visit 1.
5. AQP4-IgG is positive at visit 1 or had AQP4-IgG positive medical records before visit 1.
6. Be able to recognize English letters.
7. Patients should be on stable treatment of the following medications before screening (if anyone had a stable treatment ):

   * Immunosuppressant or immunomodulatory drugs (for example, azathioprine, cyclophosphamide, mycophenolate mofetil, tacrolimus, methotrexate and so on) must be stable for at least 8 weeks before screening and keep stable during study

     • Corticosteroids
   * At screening, the treatment dose must be stable for at least 1 month. • If patients accepted plasmapheresis or IVIg treatment, the last treatment dose/procedure must be finished at least 4 weeks ago before screening

Exclusion Criteria:

1. No acute optic neuritis and/or transverse myelitis symptoms or signs.
2. Severe NMOSD which may require plasmapheresis or intravenous immunoglobulin (IVIG) treatment, in opinion of investigator, very soon.
3. Have received plasmapheresis or IVIG treatment, the last treatment dose/procedure is less than 4 weeks before visit 1.
4. Have known autoimmune diseases other than NMOSD that would interfere with efficacy assessment or participation in this study (such as uncontrolled thyroid disease or severe rheumatoid arthritis), or have any comorbid diseases which would interfere with the efficacy evaluation of HBM9161 on NMOSD.
5. Have received rituximab or other anti-CD20 drugs treatment within 6 months before visit 1.
6. Have been used any monoclonal antibodies or research drugs for immunomodulatory effects within 3 months before visit 1 or within 5 half-life periods of the drug.
7. Females who are pregnant or lactating.
8. Patients who can't tolerate or have contraindication to high dose intravenous methylprednisolone per Investigator's opinion.
9. Have active infection at screening, or recent serious infection (i.e., requiring intravenous antimicrobial therapy or hospitalization) within 8 weeks before screening; history of or existing infection of human immunodeficiency virus(HIV), hepatitis C virus (HCV), or Mycobacterium tuberculosis. Patients must have negative test results for HCV antibody, HIV 1 and HIV 2 antibodies, and a mycobacterium tuberculosis test (test method to be determined) at visit 1.
10. Patients have positive test result for HBsAg; or HBsAg negative meanwhile HBcAb positive and HBV-DNA level>2000IU/mL.
11. Serum total IgG <700mg/dL at visit 1.
12. Absolute neutrophil count <1500个/mm3 at visit 1 and/or visit 2
13. Patients with acute liver function impairment (e.g., hepatitis) or severe liver cirrhosis (Child-Pugh Score, Class C)
14. Any malignant tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Number of treatment related adverse events (AEs) | 189 days
  Number of treatment related adverse events (AEs)

SECONDARY OUTCOMES:
Immunoglobins changes from baseline to week 27 | 189 days
  Change of concentration of immunoglobins in mg/ml overtime after administration of HBM9161 from baseline to week 27
Neurological Disability changes from baseline to week 27 | 189 days
  Neurological Disability changes from baseline to week 27 as measured by Expanded Disability Scale Score (EDSS, Score 0-10, higher means a worse outcome)
Low Contrast Visual Acuity (LCVA) changes from baseline to week 27 | 189 days
  Low Contrast Visual Acuity (LCVA) changes from baseline to week 27 as measured by Sloan Low Contrast Letter Scale (SLCLS Letter, Score 0-70, higher means a better outcome)
Patient reported improvement changes from baseline to week 27 | 189 days
  Patient reported improvement changes from baseline to week 27 as measured by Patient Global Impression-Improvement (PGI-I, Score 1-7, higher means a worse outcome)
Percentage of patients who received rescue therapy | 189 days
  Percentage of patients who received rescue therapy
Percentage of patients who have relapse | 189 days
  Percentage of patients who have relapse
Walking ability changes from baseline to week 27 | 189 days
  Walking ability changes from baseline to week 27 as measured by time used for 25-foot Walk (applicable for patients who are able to walk)
The seropositive rate of anti-HBM9161 antibody after treatment | 189 days
  Evaluation of the seropositive rate of anti-HBM9161 antibody after treatment

OTHER OUTCOMES:
Maximum change from baseline to week 27 in total serum AQP4-IgG concentrations | 189 days
  Maximum change from baseline in total serum AQP4-IgG concentrations
AQP4-IgG changes from baseline to week 27 | 189 days
  Change of serum concentration of AQP4-IgG overtime after administration of HBM9161 from baseline to week 27
HBsAb level changes from baseline to week 27 | 189 days
  Change in HBsAb level overtime after administration of HBM9161 from baseline to week 27

CONTACTS AND LOCATIONS:
Overall Officials: Wei Qiu, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Cai G, Xia S, Qin J, Liu B. Research hotspots and emerging topics in neuromyelitis optica spectrum disorder treatment: Insights from a bibliometric analysis. Medicine (Baltimore). 2025 Jun 6;104(23):e42850. doi: 10.1097/MD.0000000000042850. PMID 40489809